CLINICAL TRIAL: NCT02336321
Title: Restoration of Daily-life Hand Function Using a Brain/Neural-Computer Interaction (BNCI) System in Paralysis After Cervical Spinal Cord Injury
Brief Title: Daily-life Brain Control Of A Hand Exoskeleton After Cervical Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Institut Guttmann (Other); Scuola Superiore Sant'Anna di Studi Universitari e di Perfezionamento (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 288551-2; SO-932 (Other Grant/Funding Number: German Research Foundation (DFG)); WAY-288551 (Other Grant/Funding Number: European Commission (EC)); 01GQ0831 (Other Grant/Funding Number: Federal Ministry of Research and Education (BMBF))
Record Dates: First submitted 2014-12-19; First posted 2015-01-12 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2014-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BNCI hand-exoskeleton (Experimental): Hand motor function before, during and after application of the device
  Interventions: Device: BNCI controlled hand exoskeleton

INTERVENTIONS:
Device: BNCI controlled hand exoskeleton — The BNCI system fuses and translates bio-signals related to user intention into control signals of an assistive device performing grasping motions

SUMMARY:
In this study, 6 volunteer participants with chronic spinal cord injury will be invited to use an autonomous hand exoskeleton device controlled by a brain/neural-computer interaction (BNCI) system fusing electroencephalography (EEG) and electrooculography (EOG) to detect the intention of the user to grasp objects of daily life. The BNCI system consists of a lightweight hand exoskeleton connected to portable motors, rechargeable batteries and a computerized control system integrated into a wheelchair. Before, during and after use of the BNCI system the volunteers will perform standardized assessments and complete questionnaires to assess the functional and psychological effects of the exoskeleton. Functional outcomes primarily focus on motor function in performing daily life actions while psychological outcomes primarily focus on safety, reliability as well as predisposition and perceptions of disability.

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade A, B & C (Lower Extremity Motor Score <20)
* Motor level of injury from cervical level 4 to cervical level 7, according to ASIA guidelines
* Male and non-pregnant, non-lactating female
* Age 15-65 years old
* At least 12 months after injury

Exclusion Criteria:

* History of severe neurological injuries other than spinal cord injury (e.g. Multiple Sclerosis, Cerebral Palsy, Amyotrophic Lateral Sclerosis, Traumatic Brain Injury, Stroke)
* Concurrent medical diseases (eg. infections, circulatory, heart or lung, pressure sores) interfering with the study
* Unstable spine or unhealed limbs or pelvic fractures
* Severe spasticity (Ashworth grade 4; ie. Affected part(s) rigid in flexion or extension) or uncontrolled clonus
* Diagnosis of severe osteoporosis/penia as proven with pQCT or DXA.
* Psychiatric or cognitive conditions that may interfere with the trial
* Patients incapable of providing informed consent

Ages: 15 Years to 65 Years | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change of Toronto Rehabilitation Institute Hand Function Test (TRI-HFT) Score | Hand function will be assessed twice on the same day. Once before the hand exoskeleton is applied (absence of the assistive device) and once after the brain-controlled hand exoskeleton was attached to the patients' hand and arm.
  The TRI-HFT will be applied once before and while the patients wear the hand exoskeleton

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Guttmann, Hospital de Neurorehabilitació, Badalona, Catalonia, Spain

REFERENCES:
- [Background] Soekadar SR, Witkowski M, Vitiello N, Birbaumer N. An EEG/EOG-based hybrid brain-neural computer interaction (BNCI) system to control an exoskeleton for the paralyzed hand. Biomed Tech (Berl). 2015 Jun;60(3):199-205. doi: 10.1515/bmt-2014-0126. PMID 25490027
- [Background] Witkowski M, Cortese M, Cempini M, Mellinger J, Vitiello N, Soekadar SR. Enhancing brain-machine interface (BMI) control of a hand exoskeleton using electrooculography (EOG). J Neuroeng Rehabil. 2014 Dec 16;11:165. doi: 10.1186/1743-0003-11-165. PMID 25510922
- [Background] Cempini M, De Rossi SM, Lenzi T, Cortese M, Giovacchini F, Vitiello N, Carrozza MC. Kinematics and design of a portable and wearable exoskeleton for hand rehabilitation. IEEE Int Conf Rehabil Robot. 2013 Jun;2013:6650414. doi: 10.1109/ICORR.2013.6650414. PMID 24187233
- [Background] Cempini M, Marzegan A, Rabuffetti M, Cortese M, Vitiello N, Ferrarin M. Analysis of relative displacement between the HX wearable robotic exoskeleton and the user's hand. J Neuroeng Rehabil. 2014 Oct 18;11:147. doi: 10.1186/1743-0003-11-147. PMID 25326697